CLINICAL TRIAL: NCT06504069
Title: Effectiveness of a Virtual Reality (VR) Intervention for Prosocial Behavior and Well-being Among Adolescents: A Randomized Controlled Trial
Brief Title: A VR Intervention for Prosocial Behavior and Well-being Among Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20221208004-01
Record Dates: First submitted 2024-06-26; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-04

CONDITIONS: Adolescent

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prosocial VR Intervention (Experimental): Participants in the VR intervention group will engage in a five-week gamified prosocial VR intervention program. The intervention will consist of five weekly sessions, each lasting between 10 to 15 minutes. Each session will depict a different daily life scenario, including a home, school, street, park, and shopping mall.
  Interventions: Behavioral: Prosocial VR intervention
- Waitlist control group (No Intervention): Participants in the waitlist condition will not receive VR intervention during the study.

INTERVENTIONS:
Behavioral: Prosocial VR intervention — A five-week gamified prosocial VR intervention program based on literature review and relevance to the local contexts will be developed for the proposed project. The intervention will be expanded to include five weekly sessions, each lasting between 10 to 15 minutes. Each session will depict a different daily life scenario-home, school, street, park, and shopping mall, respectively. During each session, participants will engage in a series of tasks that incorporate elements of prosocial behavior or helping actions within the scene. These tasks are designed to be more comprehensive and interactive, ensuring that participants are fully immersed in the experience for the entire duration of the session.
  Arms: Prosocial VR Intervention

SUMMARY:
The aim of this project is to examine the effectiveness of a gamified prosocial VR intervention.

DETAILED DESCRIPTION:
There are two parts in this study. In the first part of the study, participants will be first directed to complete a background survey online (approximately 20 minutes). In the second part of the study, participants will participate in a 5-session gamified training program, one session a week for five consecutive weeks, each session lasts between 10-15 minutes. Upon completion of each session, participants will be required to complete a short 5-minute online survey. A daily diary study will be conducted during the intervention to monitor the nuance behavioral and attitudinal changes.

ELIGIBILITY:
Inclusion Criteria:

* School students aged 10-16 (i.e., primary 5 to secondary 5);
* Able to communicate in Chinese.

Exclusion Criteria:

* Significant cognitive impairment;
* Self-reported severe motion sickness;
* Uncorrected visual impairment.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Prosocial attitudes | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  Three items assessing prosocial attitudes will be revised from the Prosocial Orientation Questionnaire. Participants will rate each item on a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores on the scale indicate a greater presence of positive prosocial attitudes.
Prosocial identity | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Internalization subscale of the Self Importance of Moral Identity Scale (SIMIS) will be used to measure the construct of prosocial identity. Participants will rate each item on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Elevated scores on the scale indicate a greater degree of prosocial identity.
Prosocial intention | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Prosocial Behavioral Intentions Scale (PBIS) will be employed to evaluate individuals' future intentions to engage in prosocial behavior. Participants will rate each item on a 7-point Likert scale, ranging from 1 (Definitely would not do this) to 7 (Definitely would do this). Increased scores on the scale indicate a greater inclination towards prosocial intentions.
Attitudes toward helping others | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Attitudes toward Helping Others Scale (AHO) will be employed to assess individuals' attitudes towards helping others. Each item will be rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Elevated scores on the scale indicate a greater presence of positive attitudes towards helping others.
Altruism | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  Two items from the Preference Survey Module (PSM) will be modified to measure altruism. One example item is as follows: "Imagine the following scenario: you have won 1,000 Euros in a lottery. Considering your present circumstances, how much of the prize would you donate to a charitable cause? (Values between 0 and 1000 are permissible)." Higher scores on this item indicate a higher level of altruistic behavior or tendencies.
Empathy | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Single Item Trait Empathy Scale (SITES) will be utilized to assess levels of empathy. Participants will rate this item on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree), with higher scores indicating a greater degree of empathy.
Life satisfaction | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Satisfaction with Life Scale (SWLS) will be employed to evaluate levels of life satisfaction. Participants will rate each item on a 7-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree." Elevated scores on the scale indicate greater levels of life satisfaction.
Subjective happiness | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Subjective Happiness Scale (SHS) will be utilized to assess participants' subjective happiness. Each item will be rated on a 7-point Likert scale. Elevated scores on the scale indicate a greater level of subjective happiness.
Affect | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Emmons Mood Indicator will be employed to measure affect, encompassing two dimensions: Positive Affect and Negative Affect. Each item will be rated on a 7-point Likert scale, ranging from 1 (not at all) to 7 (extremely). Elevated scores on the scale indicate a higher level of affect.
Gratitude | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  One item from the Gratitude Adjective Checklist (GAC) will be used to measure participants' gratitude. This item will be rated on a 7-point Likert scale. A higher score indicate a higher level of gratitude.
Subjective vitality | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  Three items from the Subjective Vitality Scale (SVS) will be used to measure participants' subjective vitality. Each item will be rated on a 7-point Likert scale. Higher scores indicate a higher level of subjective vitality.
Self-esteem | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Rosenberg Self-esteem Scale (RSE) will be used to measure self-esteem. Each item will be rated on a 4-point Likert scale, ranging from 1 (strongly agree) to 4(strongly disagree). Higher scores indicate higher levels of self esteem.
Daily well-being | Daily monitoring for 5 weeks during the intervention
  Daily well-being will be assessed using a single item ("How do you feel right now?") adapted from the Well-Being Manifestations Measure Scale (WBMMS) using a sliding scale ranging from 0 (not good at all) to 100 (very good). A higher score indicates a higher level of daily well-being.
Daily prosocial act | Daily monitoring for 5 weeks during the intervention
  Daily prosocial act will be measured by one item: "How many acts have you engaged today that involve helping someone else or doing something for a good cause?" Participants will indicate the number of prosocial acts from a drop-down menu ranging from 0 to 10+. The response of "0" will be classified as "no prosocial engagement," and responses of "1" or more will be classified as "having engaged in prosocial acts."
Daily subjective happiness | Daily monitoring for 5 weeks during the intervention
  Daily subjective happiness will be measured using a condensed 2-item adaptation of the Subjective Happiness Scale (SHS). The first item will assess their self-perceived general happiness today on a scale from 1 (not at all happy) to 7 (very happy). The second item will gauge their comparative happiness to their peers during the same timeframe, ranging from 1 (less happy) to 7 (more happy). Higher scores indicate a higher level of daily subjective happiness.
Daily subjective vitality | Daily monitoring for 5 weeks during the intervention
  Daily subjective vitality will be assessed using 3 representative items from the 7-item Subjective Vitality Scale (SVS). All items will be rated on a 7-point scale (1 = not at all true to 7 = very true). Higher scores indicate a higher level of daily subjective vitality.
Daily affect | Daily monitoring for 5 weeks during the intervention
  Daily affect will be evaluated using the 9-item Emmons Mood Indicator. Participants will be instructed to rate the extent to which they experienced each emotion today using a 7-point scale (ranging from 1 = not at all to 7 = extremely). Elevated scores on the scale indicate a higher level of daily affect.
Daily gratitude | Daily monitoring for 5 weeks during the intervention
  Daily gratitude will be measured using one item from the Gratitude Adjective Checklist (GAC). This item will be rated on a 7-point Likert scale. A higher score indicates a higher level of daily gratitude.
Daily psychological needs | Daily monitoring for 5 weeks during the intervention
  Daily psychological needs will be assessed using a 9-item Basic Psychological Needs Scale (BPNS). Each subscale, namely competence, autonomy, and relatedness, consists of 3 items rated on a 7-point scale (ranging from 1 = not at all true to 7 = very true). Higher scores indicate a higher level of daily psychological needs.
Daily self-esteem | Daily monitoring for 5 weeks during the intervention
  Daily self-esteem will be evaluated using 2 items from the Rosenberg Self-Esteem Scale (Rosenberg, 1965). Ratings will be evaluated on a 4-point scale (1 = strongly disagree to 4 = strongly agree). Higher scores indicate a higher level of daily self-esteem.

SECONDARY OUTCOMES:
Intervention satisfaction | immediately after the intervention (post-intervention)
  Intervention satisfaction will be assessed using the Client Satisfaction Questionnaire-8 (CSQ-8). Participants will rate each item on a 4-point Likert scale, with "1" indicating the lowest degree of satisfaction and "4" representing the highest. Elevated scores on the scale reflect greater levels of intervention satisfaction.
Feelings in the VR | immediately after the intervention (post-intervention)
  Two items will be uesd to measure the sense of reality. Items are "I feel that the maze seemed very much like the one in the real world" and "The game scene made me feel like I was truly there".
Levels of difficulty | immediately after the intervention (post-intervention)
  Two items will be used to measure the levels of difficulty. Items are "The game is very difficult" and "The game is too difficult to operate".
Levels of interest | immediately after the intervention (post-intervention)
  Two items will be used to measure the levels of difficulty. Items are "This game is very interesting" and "I like this game".

OTHER OUTCOMES:
Socio-demographic variables | Baseline (pre-intervention)
  The study will collect socio-demographic variables including gender, age, level of education, and family income.

CONTACTS AND LOCATIONS:
Overall Officials: Bryant HUI, Ph.D., Principal Investigator — The Hong Kong Polytechnic University